CLINICAL TRIAL: NCT02463981
Title: Voluntary Anterior Insula Regulation Impacts Pain Empathy and Functional Connectivity: a Real-time fMRI Study
Brief Title: Anterior Insula Regulation and Pain Empathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Shuxia Yao, PhD student, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UESTC-SCAN-02
Record Dates: First submitted 2015-05-29; First posted 2015-06-08 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Anterior Insula Activity During Regulation; Empathic Responses After Anterior Insula Regulation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- neurofeedback training (Experimental): Neurofeedback training group receives neurofeedback from their own anterior insula.
  Interventions: Device: real-time fMRI neurofeedback training running on Turbo Brain voyager (TBV) 3.2 (Brain Innovation, Maastricht, The Netherlands)
- sham control (Sham Comparator): Sham control group receives sham neurofeedback from a large control brain region.
  Interventions: Device: real-time fMRI neurofeedback training running on Turbo Brain voyager (TBV) 3.2 (Brain Innovation, Maastricht, The Netherlands)

INTERVENTIONS:
Device: real-time fMRI neurofeedback training running on Turbo Brain voyager (TBV) 3.2 (Brain Innovation, Maastricht, The Netherlands)

SUMMARY:
The aim is to test whether rtfMRI-based neurofeedback training on anterior insula impacts pain empathy.

DETAILED DESCRIPTION:
In the present study, investigators plan to use the real-time fMRI neurofeedback to train healthy subjects to learn volitional control over their own anterior insula (AI) activity. Then the effect of AI regulation will assessed by examining subjects' empathic responses and functional connectivity changes. Subjects were separated into two groups randomly. While the experimental group received specific neurofeedback from their own AI, the control group received sham NF from an unspecific region.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury;
* claustrophobia;
* pregnancy;
* medical or psychiatric illness.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, Dr., Principal Investigator — University of Electronic Science and Technology of China

RESULTS

PARTICIPANT FLOW:
Groups:
- Neurofeedback Training: Neurofeedback training group receives neurofeedback from their own anterior insula.
  real-time fMRI neurofeedback training running on Turbo Brain voyager (TBV) 3.2 (Brain Innovation, Maastricht, The Netherlands)
- Sham Control: Sham control group receives sham neurofeedback from a large control brain region.
  real-time fMRI neurofeedback training running on Turbo Brain voyager (TBV) 3.2 (Brain Innovation, Maastricht, The Netherlands)
Period: Overall Study
Arm/Group | Neurofeedback Training | Sham Control
Started | 21 | 16
Completed | 18 | 14
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neurofeedback Training | Sham Control | Total
Number analyzed (Participants) | 21 | 16 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.2 (0.3) | 21.7 (0.5) | 21.95 (0.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 10 | 9 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  China | 21 | 16 | 37

OUTCOME MEASURES:

1. Primary Outcome: Neural Activity of Anterior Insula During Neorofeedback Training
Description: Neural activity was analyzed using standard fMRI analysis procedure that examine neural activity during training of anterior insula regulation. The measures include BOLD signal analysis (reflecting neural activity strengths) as well as functional connectivity analysis (that examine the interaction between different brain regions).
Time Frame: three days.
Population: From the initial population of 37 participants 5 had to be excluded because of high head movement during fMRI acquisition. This is a standard procedure in fMRI studies given that the analysis is very susceptible to movement artifacts.
Measure: Mean (Standard Error); unit: percentage of BOLD signal change
Arm/Group | Neurofeedback Training | Sham Control
Number analyzed (Participants) | 18 | 14
percentage of BOLD signal change | 0.077 (0.016) | 0.026 (0.018)

2. Primary Outcome: Pain Empathy Rating Scores
Description: Subjects were required to rate their empathic feeling towards painful pictures on a Likert Scale ranging from 1-9 (1 = not at all and 9 = very painful). The effects of training on the empathy for pain were analyzed comparing the feedback group with the controls group. For each subject differences were calculated between pictures that were preceded by a training compared to a no-training block. Within the context of the present design we expected that training-induced increases in anterior insula activity should lead to higher pain empathy ratings in the training group as compared to the control group.
Time Frame: three days.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Neurofeedback Training | Sham Control
Number analyzed (Participants) | 18 | 14
units on a scale | 0.249 (0.107) | -0.09 (0.122)

ADVERSE EVENTS:
Time Frame: three days - subjects were required to come back to the lab after two days.
Groups:
- Neurofeedback Training: Subjects in this group received fMRI-based feedback from their insula activity
- Sham Control: Subjects in this group received fMRI-based feedback from a unspecific control region
Arm/Group | Neurofeedback Training | Sham Control
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/16
Other Adverse Events (participants affected / at risk) | 0/21 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No